CLINICAL TRIAL: NCT00626561
Title: A Phase II Evaluation of Bevacizumab and Paclitaxel in Patients With Recurrent Small Cell, Large Cell, and Neuroendocrine Tumors of the Cervix and Uterus
Brief Title: Bevacizumab and Paclitaxel for Neuroendocrine Tumors of the Cervix
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0324
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2014-07-07 (Estimated); Last update posted 2014-07-07 (Estimated); Status verified 2014-06

CONDITIONS: Cervical Cancer; Uterine Cancer
Keywords: Cervical Cancer; Uterine Cancer; Bevacizumab; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Paclitaxel; Taxol
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Paclitaxel (Experimental): Bevacizumab 10 mg/kg intravenous (IV) twice weekly and Paclitaxel 60 mg/m^2 IV weekly.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg IV twice weekly on days 1 and 15.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Paclitaxel — 60 mg/m^2 IV weekly on days 1, 8, 15, and 22.
  Other Names: Taxol

SUMMARY:
Objectives:

Primary:

To estimate the efficacy of bevacizumab and paclitaxel in patients with recurrent small cell, large cell, and neuroendocrine cervical and uterine cancers, as measured by progression-free survival.

Secondary:

1. To estimate the efficacy of bevacizumab and paclitaxel in patients with recurrent small cell, large cell, and neuroendocrine cervical and uterine cancers, as measured by overall survival.
2. To determine the response rates in patients with recurrent small cell, large cell, and neuroendocrine cervical and uterine cancers when treated with bevacizumab and paclitaxel.
3. To characterize the quality of life (QoL) in patients with recurrent small cell, large cell, and neuroendocrine cervical and uterine cancers when treated with bevacizumab and paclitaxel.
4. To determine the nature and degree of toxicity in patients with advanced or recurrent small cell, large cell, or neuroendocrine cervical and uterine cancers when treated with bevacizumab and paclitaxel.

DETAILED DESCRIPTION:
The Study Drugs:

Paclitaxel is designed to block the mechanisms of cell division in cancer cells, which may cause them to die.

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the effects of Vascular endothelial growth factor (VEGF), a blood-vessel stimulating agent that plays an important role in the growth of both normal and abnormal blood vessels.

Study Drug Administration:

If you are found to be eligible to take part in this study, on Days 1, 8, 15, and 22 of each 28-day study "cycle", you will receive paclitaxel through a needle into your vein over 1 hour.

On Days 1 and 15 of each cycle, you will receive bevacizumab by vein. The first dose of bevacizumab will be given over about 90 minutes. If the first dose is well tolerated, the second dose may be given over about 60 minutes. If this is well tolerated, the third and any other doses may be given over about 30 minutes.

Before you receive the study drugs, you will receive premedication (selected by your doctor) to help prevent or lessen any side effects from the study drugs.

Study Visits:

About every 4 weeks, the following tests and procedures will be performed:

* You will have a physical exam, including a pelvic exam and measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 2-3 teaspoons) will be drawn for routine tests and to test how your blood clots.
* You will be asked if you have experienced any side effects.

About every 8 weeks, you will have a chest x-ray and a computed tomography (CT) or magnetic resonance imaging (MRI) scan of your abdomen and pelvis to check the status of the disease.

Length of Study:

You may stay on study for as long as you are benefitting. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

After you go off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including a pelvic exam and measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 2-3 teaspoons) will be drawn for routine tests and possibly blood clotting tests.
* You will have a CT or MRI of the abdomen and pelvis to check the status of the disease.
* You will be asked if you have experienced any side effects.

This is an investigational study. Paclitaxel is FDA approved and commercially available for the treatment of breast cancer, nonsmall cell lung cancer, ovarian cancers, and treatment of AIDS-related Kaposi's sarcoma (KS). Bevacizumab is FDA approved and commercially available for use in combination with chemotherapy in patients with colon cancer, but its use in this combination for this type of cancer is considered experimental.

Up to 20 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, advanced stage (stage IVB), recurrent, or persistent small cell, large cell, or neuroendocrine tumor of the uterine corpus and cervix
2. All patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be > / = 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or > / = 10 mm when measured by spiral CT. Biopsy confirmation is required if the lesion measures < 30 mm or if the treating physician determines it is clinically indicated.
3. Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by Response Evaluation Criteria in Solid Tumors (RECIST). Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
4. Patients must have adequate: BONE MARROW FUNCTION: Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl and platelets greater than or equal to 100,000/mcl. RENAL FUNCTION: Creatinine less than or equal to 1.5 * institutional upper limit normal (ULN), and measured or estimated creatinine clearance greater than or equal to 50 ml/min. For the purpose of estimating the creatinine clearance, the formula of Jelliffe should be utilized. HEPATIC FUNCTION: Bilirubin less than or equal to 1.5 * ULN. serum glutamate oxaloacetate transaminase (SGOT) and alkaline phosphatase less than or equal to 2.5 * ULN
5. Patients must have adequate: BLOOD COAGULATION PARAMETERS: prothrombin time (PT) such that international normalized ratio (INR) is < / = 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) < 1.2 times the upper limit of normal. NEUROLOGIC FUNCTION: Neuropathy (sensory and motor) less than or equal to [1] Common Toxicity Criteria for Adverse Effects (CTCAE) grade 1.
6. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
7. Patients with Eastern Cooperative Oncology Group (ECOG) Performance Grade of 0 or 1
8. Patients must be free of clinically significant infection.

Exclusion Criteria:

1. Patients who have progressed through or recurred within 3 months of treatment with a taxane agent administered on a weekly basis.
2. Patients who have previously been treated with bevacizumab or other anti-angiogenic agents
3. Patients who are less than 4 weeks from prior chemotherapy and/or radiation therapy
4. Patients with ECOG Performance Grade of 2, 3 or 4
5. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last 5 years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
6. Subjects meeting any of the following criteria are ineligible for study entry: (a) Inability to comply with study and/or follow-up procedures (b) Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
7. Inadequately controlled hypertension (defined as systolic blood pressure >140 or diastolic blood pressure > 90 mmHg on antihypertensive medications)
8. Any prior history of hypertensive crisis or hypertensive encephalopathy
9. New York Heart Association (NYHA) Grade II or greater congestive heart failure
10. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
11. History of stroke or transient ischemic attack within 6 months prior to study enrollment
12. Known metastatic cervical cancer to the central nervous system
13. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
14. Symptomatic peripheral vascular disease
15. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
16. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
17. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
18. Serious, non-healing wound, ulcer, or bone fracture
19. Proteinuria at screening as demonstrated by urine dipstick for proteinuria > / = 2+ (patients discovered to have > / = 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate < / = 1g of protein in 24 hours to be eligible)
20. Known hypersensitivity to any component of bevacizumab
21. Pregnant (positive pregnancy test) or lactating
22. Patients receiving black cohosh, dong quai, valerian, St. John's wort, kava kava, gotu kola. Patient cannot have received these medications within 14 days of therapy start.
23. Patients with a known hypersensitivity to taxanes, Cremophor EL (polyoxyethylated castor oil), or any component of the formulation.
24. History of hemoptysis (>/= ½ teaspoon of bright red blood per episode) within 1 month prior to Day 1
25. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 18, 2008 to November 04, 2010. All recruitment done at University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated early due to low accrual. One participant enrolled of four withdrew before being treatment.
Period: Overall Study
Arm/Group | Bevacizumab + Paclitaxel
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Population: One participant not treated.
Arm/Group | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 33 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-Free Survival is the period from study entry until disease progression, death or date of last contact.
Time Frame: Baseline to 6 Months, or until disease progression.
Population: Interim analysis was to be done after 10 patients enrolled, accrual not met. Study halted early.
Arm/Group | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data obtained every cycle (approximately every 4 weeks) until 30 days post treatment. Overall study period 2 years, May 2008 to May 2010.
Description: One participant of four was enrolled but not treated therefore excluded from adverse event reporting.
Arm/Group | Bevacizumab + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel (N=3)
Constipation (Gastrointestinal disorders) | 2
Pain (General disorders) | 2
Fatigue (General disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No